CLINICAL TRIAL: NCT05287932
Title: A Pilot Randomised Controlled Trial of a Brief Physical Activity Intervention in Older People With Multimorbidity
Brief Title: Brief Physical Activity Intervention for Older People With Multimorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Garry Tew, Professor Garry Tew, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLSGT030322
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Chronic Conditions, Multiple; Old Age; Debility; Physical Inactivity
Keywords: Multimorbidity; Older people; Physical activity
MeSH Terms: conditions — Multiple Chronic Conditions; Frailty; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Pilot randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group allocation, and participants will be asked to not disclose their allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Brief physical activity intervention including an initial 45-minute physical activity consultation, telephone support after 2 weeks (approx. 15-minute call), and provision of a pedometer, written information, and a physical activity diary. Embedded behaviour change techniques will include goal setting, self-monitoring, building self-efficacy and social support, and overcoming barriers.
  Interventions: Behavioral: Brief physical activity intervention
- Wait-list control (No Intervention): The control group will not receive any active or placebo intervention during the 4-week study period. They will also not receive any trial contacts during this period. They will however continue to be able to access their usual care from primary, secondary, community, and social services. After the final (4-week) follow-up assessment, this group will receive the full physical activity intervention.

INTERVENTIONS:
Behavioral: Brief physical activity intervention — See arm/group descriptions
  Arms: Intervention

SUMMARY:
Physical activity is an important determinant of health and well-being in older people. However, many older people do not achieve recommended physical activity levels and increasing older people's physical activity is challenging. This preliminary study will explore the effects of a brief physical activity intervention on physical activity and physical function in older people with multimorbidity. The findings will be used to inform the design of a subsequent adequately-powered randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥60 years
* 2 or more chronic conditions
* able to walk outside the home
* able to attend the study visits

Exclusion Criteria:

* living in a residential or nursing home
* housebound
* ≥3 falls in previous year
* dementia or significant cognitive impairment (unable to follow simple instructions)
* contraindication to increasing physical activity
* unable to read or speak English
* unable to provide consent
* no more than one person per household

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Average daily acceleration | 4 weeks
  Average acceleration from wrist accelerometry

SECONDARY OUTCOMES:
Intensity gradient | 4 weeks
  Intensity gradient from wrist accelerometry
Time in MVPA | 4 weeks
  Average daily time spent in moderate-to-vigorous physical activity from wrist accelerometry
Steps | 4 weeks
  Average daily step count
Muscle strengthening exercise | 4 weeks
  Average daily time spent doing muscle strengthening exercise
30-second chair rise performance | 4 weeks
  Number of sit-to-stand movements completed within 30 seconds
Handgrip strength | 4 weeks
  Maximum handgrip strength measured on both hands using a Jamar handgrip dynamometer
Timed 8ft up and go performance | 4 weeks
  Time to complete 8ft up and go test
Timed single-leg balance performance | 4 weeks
  Time able to stand on one limb
6-minute walk test performance | 4 weeks
  Total distance walked during 6-minute corridor walking test

CONTACTS AND LOCATIONS:
Overall Officials: Garry A Tew, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
External requests for this data will be considered by the Chief Investigator after the publication of the main trial findings.